CLINICAL TRIAL: NCT06621966
Title: Effectiveness of Topical Application of Olive Oil in Preventing Pressure Injuries Among Hospitalized Patients With Mobility Limitations: A Cluster Randomized Trial in the United Arab Emirates
Brief Title: Effectiveness of Topical Application of Olive Oil in Preventing Pressure Injuries
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: RAK Medical and Health Sciences University (Other)
Responsible Party: Principal Investigator, Mona Gamal, Assistant Professor, RAK Medical and Health Sciences University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAKMHSU-REC-109-2021/2022-PG-N
Record Dates: First submitted 2024-09-30; First posted 2024-10-01 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Disability Physical
Keywords: Olive oil, Pressure injury, mobility limitations, United Arab Emirates
MeSH Terms: conditions — Pressure Ulcer; Mobility Limitation | interventions — Olive Oil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental (Experimental)
  Interventions: Other: Olive Oil Topical Oil

INTERVENTIONS:
Other: Olive Oil Topical Oil — The IVG will receive standard PI prevention care along with a topical application of olive oil for 7 consecutive days. PI point prevalence and baseline risk assessments will be performed prior to the intervention. Post-intervention assessments will be conducted from days 3 to 8. Descriptive statistics and paired sample t-tests will be utilized for data analysis.

SUMMARY:
Pressure injuries (PIs) pose significant public health concerns, particularly for hospitalized patients with limited mobility. They are one of the five most common causes of harm in healthcare settings, with a global prevalence ranging from 0% to 72.5%. Hospitalized patients face a higher risk of developing PIs compared to those in community settings, with older adults (over 65 years) being particularly vulnerable.

Meta-analysis reveals a global prevalence of PIs at 14.8%, varying significantly across care settings. For instance, in acute care environments, the prevalence ranges from 6% to 18%, highlighting the need for improved preventive measures. A study in the UAE demonstrated that implementing a new intervention protocol reduced the prevalence of PIs from 2% in 2013 to 1.8% in 2018, underscoring that prevention is less costly than treatment.

Furthermore, research indicates that maintaining skin integrity is crucial in preventing PIs, with the Agency for Healthcare Research and Quality emphasizing the use of "Care Bundles" that include comprehensive skin assessments. Topical emollients and products containing hyper-oxygenated fatty acids (HOFAs) are recommended for enhancing skin hydration and reducing PI risk.

Evidence from studies in Gulf countries shows the effectiveness of olive oil in preventing and treating PIs. Despite existing interventions, recent data from the hospital conducting this study revealed a rising incidence of PIs, from 40 cases in 2020 to 55 cases in 2021. This research aims to evaluate the effectiveness of applying extra virgin olive oil topically, alongside standard preventive measures, to reduce the risk of PIs in mobility-compromised patients.

ELIGIBILITY:
Inclusion Criteria:

- mobility-limited stroke, spinal cord injuries, fractures, multiple sclerosis

Exclusion Criteria:

unwilling to participate,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change Pressure Ulcer incidence at 6 Months | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- RAKMHSU, Ras al-Khaimah, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/